CLINICAL TRIAL: NCT02608463
Title: Neuropathic Pain in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 204737
Record Dates: First submitted 2015-11-13; First posted 2015-11-18 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-05

CONDITIONS: Pain; Pregnancy
Keywords: neuropathic pain; pregnancy
MeSH Terms: conditions — Pain; Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects will participate in Part A, receive standard of care and complete the painDETECT Questionnaire (PDQ) to be assigned to 1 of 3 groups based on the PDQ score.
  Subjects in Part A will complete the following at study entry and each study visit: the Beck Depression Inventory (BDI), Visual Analogue Scale (VAS), Pain Catastrophizing Scale (PCS), and measures of pain intensity, interference, behavior. At each visit after study entry, subjects will complete the Patients' Global Impression of Change scale (PGIC); clinicians will complete the Clinical Global Impression-Global Improvement scale (CGI-I).
  Subjects in Part B will receive rTMS and be followed daily until day 29 after last rTMS session. For each session, subjects will complete a VAS prior, immediately after, and 60 minutes post, day 22 & day 29; a BDI on Days 1, 5, 12, 22, & 29; on days 5, 12, 22, & 29 subjects will complete the PGIC; clinicians will complete the CGI-I.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Part A - Neuropathic Pain (Other): Subjects with a score of ≥ 13 on the painDETECT Questionnaire (PDQ) will be assigned to the Neuropathic Pain group.
  Interventions: Behavioral: painDETECT Questionnaire; Behavioral: Pain Catastrophizing Scale; Behavioral: Pain Intensity Scale, Pain Interference Scale, Pain Behavior Scale; Behavioral: Beck Depression Inventory; Behavioral: Visual Analogue Scale; Behavioral: Patient's Global Impression of Change Scale & Clinical Global Impression-Global Improvement Scale
- Part A - Non-Neuropathic Pain (Other): Subjects with a score of ≥ 1 or ≤ 12 on the painDETECT Questionnaire (PDQ) will be assigned to the Non-Neuropathic Pain group.
  Interventions: Behavioral: painDETECT Questionnaire; Behavioral: Pain Catastrophizing Scale; Behavioral: Pain Intensity Scale, Pain Interference Scale, Pain Behavior Scale; Behavioral: Beck Depression Inventory; Behavioral: Visual Analogue Scale; Behavioral: Patient's Global Impression of Change Scale & Clinical Global Impression-Global Improvement Scale
- Part A - Control (Other): Subjects with a score of score = 0 on the painDETECT Questionnaire (PDQ) will be assigned to the Control group.
  Interventions: Behavioral: painDETECT Questionnaire; Behavioral: Pain Catastrophizing Scale; Behavioral: Pain Intensity Scale, Pain Interference Scale, Pain Behavior Scale; Behavioral: Beck Depression Inventory; Behavioral: Visual Analogue Scale; Behavioral: Patient's Global Impression of Change Scale & Clinical Global Impression-Global Improvement Scale
- Part B - rTMS (Experimental): Subjects from the Neuropathic Pain group will be invited to participate in the Part B rTMS group to receive repetitive transcranial magnetic stimulation (rTMS).
  Interventions: Behavioral: Beck Depression Inventory; Behavioral: Visual Analogue Scale; Behavioral: Patient's Global Impression of Change Scale & Clinical Global Impression-Global Improvement Scale; Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: painDETECT Questionnaire — This self-report questionnaire consists of 7 questions that address the quality of neuropathic pain syndromes. The first 5 questions ask about the gradation of pain, question 6 asks about the pain course pattern and question 7 asks about radiating pain. There are 4 additional questions (not counted in the total score) which asks the subject to rate their pain now and over the last 4 weeks and to mark on a body chart if there is pain radiating into other parts of the body.
  Other Names: PDQ
  Arms: Part A - Control; Part A - Neuropathic Pain; Part A - Non-Neuropathic Pain
Behavioral: Pain Catastrophizing Scale — The PCS is a 13-item self-report scale. It asks subjects to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification, and helplessness.
  Other Names: PCS
  Arms: Part A - Control; Part A - Neuropathic Pain; Part A - Non-Neuropathic Pain
Behavioral: Pain Intensity Scale, Pain Interference Scale, Pain Behavior Scale — The 3-item, self-report Pain Intensity assesses how much a person hurts. The first 2 items assess pain intensity over the past 7 days; the last item asks subject to rate pain intensity "right now." The 4-item, self-report Pain Interference measures the consequences of pain on relevant aspects of subject's life. It includes impairment in subject's social, cognitive, emotional, physical, & recreational activities. It also incorporates items about sleep and enjoyment of life. It assesses pain interference over the past 7 days.
  The 7-item, self-report Pain Behavior measures behaviors that typically indicate to others that an individual is experiencing pain. Measures include observations (sighing, crying), behaviors (resting, guarding, facial expressions, asking for help), & verbal reports of pain. It assesses pain interference over the past 7 days.
  All three scales, derived from the Patient Reported Outcomes Measurement Information System (PROMIS), are not disease specific.
  Other Names: Pain Measures
  Arms: Part A - Control; Part A - Neuropathic Pain; Part A - Non-Neuropathic Pain
Behavioral: Beck Depression Inventory — The BDI is a widely used instrument that has been used in both clinical and non-clinical setting measuring depressive symptoms. It is a 21 item questionnaire with 4-5 responses for each question. Responses are coded 0-3 for the 4 point scales. The 5 point scales include an additional 2a and 2b response code. The symptom categories reflect overt behavioral manifestations of depression. The instrument has both a high degree of reliability and validity (Beck, Ward, Mendelson, Mock & Erbaugh, 1961).
  Other Names: BDI
Behavioral: Visual Analogue Scale — 100 mm line scale that is subject administered to subjectively rate current pain symptoms. The subject will be instructed to draw a single vertical line that best describes current state.
  Other Names: VAS
Behavioral: Patient's Global Impression of Change Scale & Clinical Global Impression-Global Improvement Scale — The PGIC gives a global rating of change in symptoms, activities, emotion, and overall quality of life related to the subject's pain condition. This is a self-rated scale.
  The CGI-I gives a global rating of the improvement/change in the symptoms since the last study visit. This is administered by the MD.
  Other Names: PGIC & CGI-I
Device: Transcranial Magnetic Stimulation — Subjects will undergo daily repetitive transcranial magnetic stimulation (rTMS), defined as Monday through Friday, for a total of 10 consecutive sessions. rTMS will be applied using the NeuroStar TMS Therapy System through a figure-8 coil connected to a magnetic stimulator, which provides a biphasic pulse. The coil is applied to the primary motor cortex, M1, contralateral to the painful side. The optimal stimulus site, motor hot spot, will be determined according to visual detection of muscle twitches, and a resting motor threshold is defined as the minimal intensity necessary to induce at least one visible muscle twitch. An rTMS session consists of 10 trains at 90% intensity of resting motor threshold (one train, 100 pulses at 10 Hz; intertrain interval, 50s).
  Other Names: NeuroStar® TMS
  Arms: Part B - rTMS

SUMMARY:
This will be the first study to investigate the use of rTMS in the treatment of neuropathic pain in pregnancy. This study will enroll 60 pregnant subjects, age 18-45. All participants will receive treatment as usual. Subjects diagnosed with neuropathic pain will be offered rTMS as a treatment option.

DETAILED DESCRIPTION:
Neuropathic pain is a common pain disorder that is caused by problems in the nervous system. It affects more women than men and commonly occurs in pregnancy. Physicians have little information to guide their treatment of neuropathic pain in pregnancy. The overall goal of this study is to define the course, management, and pregnancy outcomes of neuropathic pain in pregnancy and the acute postpartum period. It is difficult to manage neuropathic pain in pregnancy as treatment options must minimize their risk to the unborn child as they have a direct effect on infant outcomes through their exposure in utero. Thus, other treatments are needed. Repetitive transcranial magnetic stimulation (rTMS) may be an acceptable alternative to medications. Transcranial magnetic stimulation uses a magnetic force to change the way nerves work in the brain. This non-invasive and localized mechanism of action makes it attractive for use in special populations, such as pregnancy. Study visits will occur approximately every 4-6 weeks during pregnancy until approximately 3 months postpartum for a maximum of 12 visits.

ELIGIBILITY:
Part A

Inclusion Criteria:

* age 18-45 years old,
* ability to give informed consent,
* viable pregnancy, and
* enrollment prior or equal to 24 weeks gestation

Exclusion Criteria:

* Active or history of substance use disorder within the past year
* Non-English speaking

Part B

Inclusion Criteria:

* Subjects enrolled in Part A and willing to consent to Part B of this protocol
* Pregnant with current chronic neuropathic pain
* Subjects failed treatment with amitriptyline or nortriptyline as defined by one of the following:

  * no clinical improvement following a 4-week trial of amitriptyline or nortriptyline (i.e., CGI-I score ≥4)
  * an inability to tolerate the medication (i.e., side effects)
* Subjects must pass the TMS Safety Checklist Adult Safety Screen (TASS).
* Subjects should be off medication, which can lower seizure thresholds (e.g., amitriptyline and nortriptyline) for at least two weeks prior to study entry.
* Subjects with neuropathic pain including those with diagnosis of spinal cord injury, fibromyalgia, compression neuropathies (including diabetic peripheral neuropathy), post stroke pain, and multiple sclerosis
* Subjects with a baseline VAS score greater than 30

Exclusion Criteria:

* Current or past history of a seizure disorder (e.g., epilepsy)
* Current history of preeclampsia
* Current or history of brain lesions (e.g., aneurysm)
* History of major head trauma (e.g., stroke; previous cranial neurosurgery)
* Ferromagnetic metal in the head, neck, or chest (e.g., plates or pins, bullets, shrapnel)
* Microprocessor implants in the head (e.g., cochlear implants) or life-sustaining microprocessor implants anywhere in the body (e.g., prosthetic cardiac valves)
* Cardiac pacemaker
* Active or inactive implants (e.g., deep brain stimulators, vagus nerve stimulators)
* Active treatment with medications that lower seizure threshold (e.g., bupropion, amitriptyline, nortriptyline, or other TCA)
* Increased intracranial pressure (which lowers seizure threshold)
* Implanted medication pumps
* Intracardiac lines
* Significant heart disease defined as heart disease that causes moderate to severe symptoms and/or is characterized by moderate to severe pathology, including a recent history of myocardial infarction and heart failure with an ejection fraction of less than 30% or with a New York Heart Association Functional Classification of Class III or IV.
* Bipolar disorder (to reduce the risk of mania)
* History of suicide attempt(s)
* Family history of epilepsy
* Heavy alcohol consumption within the past 48 hours
* Permanent makeup or tattoos with metallic dyes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shona L Ray-Grififth, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Neuropathic Pain Group: ≥13 on the painDETECT Questionnaire (PDQ) 10 subjects
- Part A: Non-Neuropathic Pain Group: ≥1 and ≤12 on the PDQ 5 subjects
- Part A: Controls: Patients without neuropathic pain receiving care as usual.
- Part B Participants: No participants were ever enrolled in Part B, so this group has been dropped from all future sections.
Period: Overall Study
Arm/Group | Part A: Neuropathic Pain Group | Part A: Non-Neuropathic Pain Group | Part A: Controls | Part B Participants
Started | 10 | 5 | 0 | 0 (No study participants were enrolled in Part B.)
Completed | 10 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 subjects met criteria to be assigned to the "control" group
Groups:
- Neuropathic Pain Group: ≥13 on the painDETECT Questionnaire (PDQ)
- Non-Neuropathic Pain Group: score of ≥1 or ≤12 on the PDQ
- Controls: Patients without neuropathic pain receiving care as usual.
- Total: Total of all reporting groups
Arm/Group | Neuropathic Pain Group | Non-Neuropathic Pain Group | Controls | Total
Number analyzed (Participants) | 10 | 5 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 0 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 29.4 [24 to 37] | 29.4 [24 to 36] |  | 29.4 [24 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 0 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 0 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 4 | 0 | 14
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Analogue Scale for Pain
Description: 100 mm line scale that is subject administered to subjectively rate current pain symptoms. The subject will be instructed to draw a single vertical line that best describes current state. The total score ranges from 0-100 with higher numbers indicating worse outcomes. The VAS will be administered at every subject visit.
Time Frame: Baseline and end of study participation, an average of 194 days
Population: No subjects were ever assigned to the control group, so no stats were performed on this group
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Neuropathic Pain Group: ≥13 on the painDETECT Questionnaire (PDQ) 10 subjects
- Non-Neuropathic Pain Group: ≥1 and ≤12 on the PDQ 5 subjects
- Control: Patients without neuropathic pain receiving care as usual. Due to n=0, no statistical analysis was completed.
Arm/Group | Neuropathic Pain Group | Non-Neuropathic Pain Group | Control
Number analyzed (Participants) | 10 | 5 | 0
score on a scale | -0.57 [-18.26 to 17.12] | -14.4 [-47.02 to 18.22] |

ADVERSE EVENTS:
Time Frame: Average length of study participation: 194 days; Range: 112-259 days
Description: None of the subjects met criteria to be assigned to the "control" group
Groups:
- Neuropathic Pain Group: score of ≥13 on the PDQ
  Total Serious Adverse Events: 6 Number of Participants Affected by Serious Adverse Events: 3
  Total Adverse Events: 62 Number of Participants Affected by Adverse Events: 8
- Non-Neuropathic Pain Group: score of ≥ 1 or ≤ 12 on the PDQ
  Total Serious Adverse Events: 40 Number of Participants Affected by Serious Adverse Events: 3
  Total Adverse Events: 39 Number of Participants Affected by Adverse Events: 5
- Controls: score of 0 on the PDQ
  Total Serious Adverse Events: 0 Number of Participants Affected by Serious Adverse Events: 0
  Total Adverse Events: 0 Number of Participants Affected by Adverse Events: 0
Arm/Group | Neuropathic Pain Group | Non-Neuropathic Pain Group | Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/10 | 3/5 | 0/0
Other Adverse Events (participants affected / at risk) | 8/10 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuropathic Pain Group (N=10) | Non-Neuropathic Pain Group (N=5) | Controls (N=0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 — Intubated, ventilator support, NICU
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 — Glucose given, NICU
Patent Ductus Arteriosus (Cardiac disorders) | 0 (0) | 1 (1) | 0 — Admitted to NICU, given ECHO
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 — Start date: 8/28/2019 End date: Ongoing 4 - Unrelated to Study Device 5- Intervention Phototherapy
Severe Retro-Micrognathia with Critical Airway (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5- Intervention Tracheotomy
Microtia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Intervention CT Scan & Hearing evaluations
Microstomia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Placed gastrostomy tube & CT Scan
Vertebral Anomalies (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Chest X-Rays & consulted orthopedics
Infection of Tracheotomy (Infections and infestations) | 0 (0) | 1 (1) | 0 — Start Date: 09/24/2017 End Date: 9/30/2017 4 - Unrelated to Study Device 5 - antibiotics & culture
Acinetobacter Infection of GT site (Infections and infestations) | 0 (0) | 1 (1) | 0 — Start Date: 10/20/2017 End Date: 10/30/2017 4 - Unrelated to Study Device 5 - cultured infection & antibiotics
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - placed gastrostomy tube & speech therapy evaluation
Cleft Palate (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - discovered 5/4/2018 in clinical exam
Bilateral superior vena cava without bridging vein (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - admitted to NICU & given ECHO
Shortened Femurs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing
Bilateral Club Feet (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 1 - discovered in clinical exam
Teratologic Hips (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 — Start Date: 9/1/2017 End Date: Ongoing 4 - Unrelated to Study Device 1 - discovered by abdominal x-ray
Glossoptosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 — Start Date: 8/28/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - gastrostomy feeding tube
Medical neglect of child by caregiver (Social circumstances) | 0 (0) | 1 (1) | 0 — Start Date: 11/21/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - DHS Report
Cardiopulmonary arrest with successful resuscitation (Cardiac disorders) | 0 (0) | 2 (2) | 0 — Start Date: 12/06/2017 End Date: 12/06/2017 4 - Unrelated to Study Device 5 - CPR
Moraxella catarrhalis & HFLU Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 — Start Date: 12/04/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Culture & antibiotics
Hypochloremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 — Start Date: 11/26/2017 End Date: 12/06/2017 4 - Unrelated to Study Device 5 - IV fluids & medications
Hyperactive Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 — Start Date: 11/20/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Medications for Sedation
Rhinovirus Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 — Start Date: 11/21/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - medication
Preeclampsia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 — Start Date: 11/10/2016 End Date: 11/10/2016 4 - Unrelated to Study Device 5 - Emergency C-section
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 — Start Date: 11/10/2016 End Date: 11/12/2016 4 - Unrelated to Study Device 5 - NICU Admission
Pre-Term Labor (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 — Start Date(s): 03/04/2017; 01/10/2017 End Date(s): 03/04/2017; 01/11/2017 4 - Unrelated to Study Device 5 - Emergency C-section
Incision Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 — Start Date: 03/04/2017 End Date: Ongoing 4 - Unrelated to Study Device 5 - Surgery & Wound Care
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 — Start Date: 12/08/2016 End Date: 02/16/2017 4 - Unrelated to Study Device 5 - Antibiotic, cough syrup, admission to hospital
Hellp Syndrome (Atypical) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 — Start Date: 04/15/2017 End Date: 04/20/2017 4 - Unrelated to Study Device 5 - Hospital & Nifedipine
Neonatal Abstinence Syndrome (Social circumstances) | 1 (1) | 2 (2) | 0 — Start Date(s): 04/15/2017; 04/15/2017 End Date(s): 04/29/2017; 04/29/2017 4 - Unrelated to Study Device 5 - NICU Admission
Meconium Aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 — Start Date: 04/20/2017 End Date: 04/22/2017 4 - Unrelated to Study Device 5 - NICU Admission
Transient Trachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 — Start Date: 04/20/2017 End Date: 04/22/2017
Metabolic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0
seizure-like activity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0
Preterm Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0
Patent foramen ovale (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0
Severe Retro-Micrognathia with critical airway (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuropathic Pain Group (N=10) | Non-Neuropathic Pain Group (N=5) | Controls (N=0)
Pain Increase (Nervous system disorders) | 8 | 3 | 0 (0) — Start Date(s): 10/27/2016; 12/01/2016; 11/17/2016; 12/22/2016; 02/16/2017; 11/17/2016; 07/13/2017; 12/01/2016; 12/01/2016; 04/06/201; 06/01/2017; 04/13/2017; 05/11/2017; 05/18/2017; 08/10/2017
Headaches (Nervous system disorders) | 3 | 2 | 0 (0) — Start Date(s): 11/17/2016; 06/05/2017;02/13/2017; 04/27/2017; 11/03/2016;12/01/2016; 06/01/2017; 05/18/2017; 08/03/2017 4 - Unrelated to Study Device 3 - Resolved / Recovered
Anesthesia Difficulty (Nervous system disorders) | 1 | 0 | 0 — Start Date: 12/16/2016 End Date: 12/16/2016 4 - Unrelated to study device 1 - Recovered / Resolved
Depressed Mood (Psychiatric disorders) | 4 | 2 | 0 (0) — Start Date(s): 10/27/2016; 09/22/2016; 07/13/2017; 05/26/2017; 12/01/20160; 6/01/2017; 06/08/2017; 04/13/2017; 05/18/2017; 07/13/2017; 08/10/2017f 4 - Unrelated to study device 2 - recovering / resolving
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 (0) — Start Date(s): 01/26/2017; 12/22/2016 End Date(s): Ongoing 4 - Unrelated to study device 3 - Not recovered / resolved
Dry Mouth (Blood and lymphatic system disorders) | 1 | 0 | 0 (0) — Start Date: 01/26/2017 End Date: Ongoing 4 - Unrelated to Study Device 3 - Not recovered / resolved
Dizzy Spells (Metabolism and nutrition disorders) | 1 | 0 | 0 (0) — Start Date: 02/23/2017 End Date: Ongoing 4 - Unrelated to study device 2 - Recovering / Resolving
Vision Changes (Eye disorders) | 1 | 0 | 0 (0) — Start Date: 11/17/2016 End Date: 12/16/2016 4 - Unrelated to Study Device 1- Recovered / Resolved
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 (0) — Start Date(s): 02/23/2017; 11/03/2016; 11/17/2016; 08/31/2016; 02/16/2017; 12/01/2016; 02/26/2017; 04/27/2017; 06/29/2017; 08/10/2017 4- Unrelated to Study Device 5 - Recovered Resolved
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 (0) — Start Date(s): 02/23/2017; 12/01/2016; 02/26/2017; 04/27/2017 4 - Unrelated to study device 1 - Recovered / Resolved
Insomnia (Psychiatric disorders) | 3 | 2 | 0 (0) — Start Date(s): 08/25/2016; 11/03/2016; 02/16/2017; 10/17/2016; 08/31/2016; 12/01/2016; 04/06/2017; 02/23/2017; 04/13/2017; 06/08/2017; 06/15/2017; 04/27/2017; 08/10/2017 4- Unrelated to the study device 1 - resolved / recovered
Irritability (Psychiatric disorders) | 1 | 0 | 0 (0) — Start Date(s): 08/25/2016; 08/23/2017 4 - Unrelated to the study device 1 - Recovered / Resolved
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 (0) — Start Date: 09/22/2016 End Date: Ongoing 4 - Unrelated to the study device 6 - Unknown
Braxton Hicks Contractions (Reproductive system and breast disorders) | 0 | 1 | 0 (0) — Start Date: 10/09/2016 End Date: 11/10/2016 4 - Unrelated to the study device 1- Recovered / Resolved
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 (0) — Start Date: 10/20/2016; 09/22/2016; 05/04/2017; 02/02/2017 4 - Unrelated to study device 1 - Recovered / Resolved
Carpel Tunnel (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 (0) — Start Date: 10/20/2016 End Date: Ongoing 4 - Unrelated to Study Device 3 - Not recovered / resolved
Anxiety (Psychiatric disorders) | 1 | 1 | 0 (0) — Start Date(s): 12/22/2016; 02/09/2017; 03/02/2017; 04/13/2017 4 - Unrelated to study device 3 - not recovered / resolved
Hypervigilance (Psychiatric disorders) | 0 | 1 | 0 (0) — Start Date: 01/26/2017 End Date: Ongoing 4 - Unrelated to Study Device 3 - Not recovered / resolved
Drowsiness or sedation (Psychiatric disorders) | 1 | 1 | 0 (0) — Start Date: 09/22/2016; 12/12/2016 4 - Unrelated to study device 6 - Unknown
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 (0) — Start Date: 09/22/2016 End Date: Ongoing 4 - Unrelated to study device 3 - not recovered / resolved
Vaginal Bleeding (Reproductive system and breast disorders) | 2 | 0 | 0 (0) — Start Date: 10/27/2016; 02/23/2017 End Date: 10/27/2016; 03/16/2017 4 - Unrelated to study device 1 - recovered / resolved
Bilateral Feet Edema (Blood and lymphatic system disorders) | 3 | 0 | 0 (0) — Start Date: 10/24/2016 End Date: 10/27/2016 4 - Unrelated to study device 1 - recovered / resolved
Fatigue (Psychiatric disorders) | 1 | 0 | 0 (0) — Start Date(s): 02/16/2017; 10/17/2016 End Date: Ongoing 4 - Unrelated to study device 3 - not resolved / recovered
Postpartum Depression (Psychiatric disorders) | 2 | 1 | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 | 0 | 0 (0) — Start Date(s): 11/17/2016; 11/16/2016; 06/29/2017 4 - Unrelated to Study Device 1 - Recovered / resolved
Lip Tie (General disorders) | 1 | 0 | 0 (0) — Start Date: 05/27/2017 End Date: Ongoing 4 - Unrelated to study device 4 - Residual effects present, not treated
Right Ankle Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 (0) — Start Date: 05/08/2017 End Date: 06/22/2017 4 - Unrelated to study device 1 - recovered / resolved
Allergies (Immune system disorders) | 0 | 1 | 0 (0) — Start Date(s): 08/31/2017; 04/27/2017 4 - Unrelated to study device 1 - recovered / resolved
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 (0) — Start Date: 10/26/2016; 12/21/2016; 06/29/2017; 04/13/2017 End Date: 11/02/2016; 12/28/2016; 06/29/2017; 05/24/2017 4 - Unrelated to study device 1 - resolved / recovered
Abdominal Cramps (Gastrointestinal disorders) | 0 | 1 | 0 (0) — Start Date: 05/23/2017 End Date: 07/17/2017 4 - unrelated to study device 1 - resolved / recovered
Bacterial Vaginosis (Reproductive system and breast disorders) | 0 | 1 | 0 (0) — Start Date: 02/05/2017 End Date: 02/16/2017 4 - Unrelated to study device 1 - resolved / recovered
Urinary Tract Infection (Reproductive system and breast disorders) | 0 | 1 | 0 (0) — Start Date: 02/10/2017 End Date 03/019/2017 4 - unrelated to study device 1 - resolved / recovered
Yeast Infection (Reproductive system and breast disorders) | 0 | 1 | 0 (0) — Start Date: 02/10/2017 End Date: 02/16/2017 4 - unrelated to study device 1 - resolved / recovered
Skin Burning (Injury, poisoning and procedural complications) | 0 | 1 | 0 (0) — Start Date: 05/27/2017 End Date: 05/27/2017 4 - unrelated to study device 1 - resolved / recovered
Mastitis (Reproductive system and breast disorders) | 0 | 1 | 0 (0) — Start Date: 05/26/2017 End Date: Ongoing 4 - unrelated to study device 3 - not resolved / recovered
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 (0) — Start Date: 06/29/2017 End Date: Ongoing 4 - unrelated to study device 3 - not resolved / recovered
Hemorrhoid (Gastrointestinal disorders) | 2 | 0 | 0 (0) — Start Date: 02/23/2017; 06/29/2017 End Date: Ongoing 4 - unrelated to study device 3 - not resolved / recovered
Sciatica (Nervous system disorders) | 2 | 1 | 0 (0)
Tooth pain or Absess (Gastrointestinal disorders) | 1 | 1 | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 (0)
Weight Loss (Gastrointestinal disorders) | 1 (1) | 0 | 0 (0) — Start Date: 06/29/2017 End Date: Ongoing 4 - unrelated to study device 3 - not resolved / recovered
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 (0) — Start Date: 04/13/2017 End Date: 05/11/2017 4 - unrelated to study device 1 - resolved / recovered
Weight Gain (Gastrointestinal disorders) | 1 (1) | 0 | 0 (0) — Start Date: 04/27/2017 End Date: Ongoing 4 - unrelated to study device 3 - not resolved / recovered
Hypertension (Cardiac disorders) | 2 | 1 | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 | 0 (0) — Start Date: 05/15/2017 End Date: 05/15/2017 4 - unrelated to study device 1 - resolved / recovered
Flank Pain (Renal and urinary disorders) | 1 | 0 | 0
Bilateral Hand Edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Numbness/tingling of bilateral hands (Nervous system disorders) | 1 | 0 | 0
Preterm Labor (Reproductive system and breast disorders) | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Low Lying Kidneys (Renal and urinary disorders) | 0 | 1 | 0
Cellulitis at gastrostomy tube site (Gastrointestinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination due to inability to enroll pregnant subjects into the TMS intervention portion (Part B) of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT02608463/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT02608463/SAP_003.pdf